CLINICAL TRIAL: NCT00194610
Title: Botox (Botulinum Toxin A) as a Treatment for Interstitial Cystitis in Women: A Randomized Placebo Controlled Trial
Brief Title: Botox as a Treatment for Interstitial Cystitis in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Paul G. Allen Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25398-D
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox injection (Experimental): Subjects were injected with Botulinum toxin A in a mix of 50 U diluted in 2 cubic centimeters of normal saline. With the subjects in the dorsal lithotomy position, one injection of 25 international units was given into the bladder neck at the 3 o'clock position and another of 25 international units was given into the 9 o'clock position
  Interventions: Drug: Botox
- Normal saline (Placebo Comparator): Subjects were injected in the bladder neck with 1 cubic centimeter normal saline into the 3 o'clock and 6 o' clock positions in the perineum, while in the dorsal lithotomy position
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Botox — Botox 25 international units per injection injected in two places in the bladder neck, with option to inject two other tender points with 25 units each
  Other Names: Botulinum Toxin A
  Arms: Botox injection
Other: normal saline — Normal saline injected into the bladder neck via the perineum, 1 cc each given at positions 3 o'clock and 9 o'clock
  Arms: Normal saline

SUMMARY:
Patients with interstitial cystitis have been well documented to have pelvic floor muscle tenderness as well as pain on bladder distension. Some investigators have even suggested that pelvic floor muscle pain is primarily the cause of bladder problems.

Botulinum toxin A causes muscle relaxation by inhibiting the acetylcholine release at the neuromuscular junction. It has been shown that this mechanism relieves pain in a number of muscle spasm-related syndromes.

Because, at present, there is little effective therapy available for patients with interstitial cystitis, the researchers want to determine if botulinum toxin A will relieve bladder and pelvic pain in these patients.

DETAILED DESCRIPTION:
Screening Visit:

After being screened by her medical provider, the patient will be given the opportunity to ask questions about the study. She will then be asked to read and sign the consent and then be randomized.

Then, for women of childbearing age, a pregnancy test will be done.

Next, we will ask the patient to fill out baseline study forms and she will be given a Voiding Diary. She will also be asked to provide a urine sample which will be processed for chemistry and culture.

Injection Visit:

This visit will be scheduled one week after the Screening Visit. First, a standard history and physical will be done. Then the clinician will proceed with the injection. The subject will receive an injection of not more than 5 ml of 1% lidocaine without epinephrine at the site of the botulinum toxin A injection.

Next, 25 units of Botox will be injected, via the transvaginal route, on either side of the bladder neck. The remaining 50 units will be injected (in 2 - 25 unit doses) into other pelvic sites that the patient has identified as tender during the patient examination.

1 Month Post Injection Mailing: The patient will be mailed a packet containing follow-up questionnaires and asked to mail them back upon completion.

6 Week Urine Collection Visit: Two weeks after receiving her study injection, we will ask the patient to go to the Urology Clinic and provide a urine sample.

2 Month Post Injection Mailing: Same as 1 Month Post Injection Visit.

3 Month Post Visit: The subject will be asked to fill out follow-up questionnaires and will be asked to turn in her last set of Voiding Diaries.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 and older
* Diagnosis of interstitial cystitis
* Subject has severity/stage of disease: at least 12 voids/day with the presence of pelvic pain
* Ability to follow study instructions and likely to complete all required visits.
* Negative urine pregnancy test on the day of treatment prior to the administration of study medication (for females of childbearing potential; if applicable)

Exclusion Criteria:

* Use of any medications that might interfere with neuromuscular function
* Any medical condition that may put the subject at increased risk with exposure to Botox including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study
* Known allergy or sensitivity to any of the components in the study medication
* Concurrent participation in another investigational drug or device study, or participation in the 30 days immediately prior to study enrollment.
* Stress incontinence
* Urinary tract infection at time of enrollment
* Overtly psychotic or suicidal
* Pain from another source in the genital tract such as kidney stones or neoplasm
* Having had radiation therapy
* History of genitourinary tuberculosis
* Neurological abnormalities such as stroke, brain tumors, spinal cord injury and Parkinson's or Alzheimer's disease
* Currently taking antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-05; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Yang, MD, Principal Investigator — University of Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 subjects were recruited to a double blind study comparing Botulinum toxin A to normal saline. Each subject received either 50 units of Botulinum Toxin A or normal saline in the periurethral tissue in the Urology Clinic of the University of Washington.
Pre-assignment Details: No pre-assignment criteria were used.
Groups:
- Saline: Total 2 cc injected periurethrally
- Botox: Botox 25 IU injected bilaterally periurethrally for a total of 50 IU. Possible but not mandatory was two more injections of 25 IU in each of two trigger points
Period: Overall Study
Arm/Group | Saline | Botox
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Botox | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Females | 11 | 9 | 20
  Males | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Chronic Prostatitis Symptom Index (CPSI-F)
Description: CPSI-F was adapted from the CPSI, in order to document the location of pain, with working pertinent to female anatomy. The CPSI-F was scored on a range of 0-83 (0-61 in the pain domain, 0-10 in the urination domain, 0-6 in the impact of symptoms domain, and 0-6 in the quality of life domain), with higher scores denoting worse symptoms.
Time Frame: 3 months
Population: Total number of subjects was based on clinical volume, and subjects were randomized into each of two arms.
Measure: Mean (Standard Deviation); unit: Total CPSI-F
Groups:
- Placebo : Saline: Saline 2 cc total injected periurethrally
- Experimental Intervention: Botox: Botulinum toxin 25 IU injected bilaterally periurethrally for a total of 50 IU. Possible, but not mandatory, injections of 25 IU in each of 2 trigger points.
Arm/Group | Placebo : Saline | Experimental Intervention: Botox
Number analyzed (Participants) | 11 | 9
Total CPSI-F | 29.6 (8.0) | 35.2 (3.9)

ADVERSE EVENTS:
Arm/Group | Saline | Botox
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes